CLINICAL TRIAL: NCT03060239
Title: Exploration of the Mechanism of Movement Improvement During Rapid Eye Movement (REM) Sleep Behaviour Disorder (RBD) in Parkinson's Disease Using Near-infrared Spectroscopy (NIRS)
Brief Title: Exploration of the Mechanism of Movement Improvement During RBD in Parkinson's Disease Using NIRS
Acronym: NIRS-RBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Beau Soleil (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-A01532-42
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Near infrared Spectroscopy; REM sleep behaviour disorder; Supplementary motor area
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Patients with Parkinson's disease with severe REM sleep behaviour disorder according to International Classification of Sleep Disorders (ICSD2) criteria.
  Interventions: Other: Near Infrared Spectroscopy

INTERVENTIONS:
Other: Near Infrared Spectroscopy — Use of the near-infrared-spectroscopy (NIRS) to explore the cortical mechanism by which this sleep disorder would allow a disappearance of parkinsonian signs at night

SUMMARY:
The purpose of this study is to confirm the improvement of movement during RBD in Parkinson's disease and to explore the neuronal network involved in this improvement using NIRS.

DETAILED DESCRIPTION:
The aim of this study is to compare the quality of movement during REM sleep during RBD episodes and movement awake without and with dopaminergic treatment while measuring cortical activity using NIRS.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease (Hughes AJ et al., 2001)
* Patients with REM sleep behaviour sleep disorder according to the ICSD2 (International Classification of Sleep Disorders 2) criteria and frequent reported several times per week by the spouse
* Informed written consent signed
* Patient aged 40 to 90 years
* Affiliate or benefiting from a social security scheme.

Exclusion Criteria:

* Atypical Parkinson's Syndromes
* Patient not accepting polysomnography

  * Contraindications to cerebral Magnetic Resonnance Imaging (MRI): pacemaker, cochlear implants, certain heart valves, claustrophobia, pregnancy.
  * Limit of validity of the MRI: if the patient presents dyskinesias preventing immobile maintenance of a few minutes in the MRI for the acquisition of images

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Difference of signal NIRS on the supplementary motor area (SMA) during the movement realized during the REM sleep behaviour disorder (RBD) and reproduced in standby in the patient parkinsonian in "on". | 24 hours
  Difference of signal NIRS on the supplementary motor area (SMA) during the movement realized during the REM sleep behaviour disorder (RBD) and reproduced in standby in the patient parkinsonian in "on" (means that the patient is under effective dopaminergic treatment).
  The NIRS signal corresponds to the area under curve (AUC) of the oxyhemoglobin (O2Hb) and desoxyhemoglobin concentration's variation during duration of the movement.

SECONDARY OUTCOMES:
Difference of NIRS signal in different cortical regions and in different conditions: rest, movement "on" and "off", RBD, and in standby. | 24 hours
  Difference of NIRS signal in different cortical regions and in different conditions: rest, movement "on"(means that the patient is under effective dopaminergic treatment ) and movement "off" (means that the patient has been weaned from any treatment for several hours), RBD (REM sleep behavior disorder), and in standby.
Difference of movement speed measured by accelerometers under different conditions. | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Beau Soleil, Montpellier, France